CLINICAL TRIAL: NCT03903575
Title: 3D Comparison of Anterior Teeth Retraction and Anchorage Control Between En-masse and Two-step Mechanics: A Randomized Prospective Clinical Trial
Brief Title: 3D Comparison of Anterior Teeth Retraction and Anchorage Control Between En-masse and Two-step Mechanics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Sergio Roberto de Oliveira Caetano, Masters in Orthodontics, PhD Student, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04186818.2.0000.5259
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Malocclusion, Angle Class I; Bimaxillary Protrusion; Orthodontic Space Closure
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Intervention Model Description: All 32 patients will be randomly allocated in a 1:1 ratio to either en masse (n=16) group or the two-step anterior retraction (n=16) group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- En Masse Retraction (Experimental): Group treated by retracting the six anterior teeth simultaneously.
  Interventions: Procedure: En masse anterior teeth retraction
- Two-Step Retraction (Active Comparator): Group treated by retracting the canines incisors in two different steps.
  Interventions: Procedure: Two-Step Retraction

INTERVENTIONS:
Procedure: En masse anterior teeth retraction — After extraction of the four premolars the posterior teeth will be tied-together and the six anterior teeth will be retracted by sliding mechanics.
  Arms: En Masse Retraction
Procedure: Two-Step Retraction — After extraction of the four premolars the posterior teeth will be tied-together and the canines will be retracted by sliding mechanics. After the distalization of the canines they will be tied to the posterior teeth and the incisors will be retracted by sliding mechanics.
  Arms: Two-Step Retraction

SUMMARY:
The aim of this study is to compare en masse (EM) and two-step anterior teeth retraction (TSR) evaluated by means of three-dimensional images superimposition. Thirty-two adult patients with bimaxillary protrusion planed for treatment with four first premolar extractions will be enrolled. All patients will be randomly allocated in a 1:1 ratio to either EM (n=16) group or the TSR (n=16) group. Cone bean computed tomography will be taken before and after anterior retraction. A blind observer will construct separate 3D models for maxillary and mandibular surfaces using the anterior cranial fossa to register models of before and after space closing. Quantitative assessment of posterior anchorage loss and amount of anterior teeth retraction are the main outcomes. The secondary outcomes are the inclination of the molars, canines and incisors.

ELIGIBILITY:
Inclusion Criteria:

* Angle Class I malocclusion;
* Bimaxillary protrusion;
* Convex profile;
* All natural teeth present in the mouth;
* Absence of crowding or with negative discrepancy up to 4mm;
* Absence of vertical and transverse occlusal problems;
* Good oral health;
* Good general health.

Exclusion Criteria:

* Lack of time to attend consultations;
* Patients with severe systemic and psychological illness;
* Patients with parafunction (bruxism), reflux or eating disorders;
* Presence of periodontal disease;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Anchorage loss | 12 months
  Quantitative assessment of posterior anchorage loss between the two groups as measured by tomographic superimposition at the end of space closure.
Anterior teeth retraction | 12 months
  Quantitative assessment of anterior teeth retraction between the two groups as measured by tomographic superimposition at the end of space closure.

SECONDARY OUTCOMES:
Molar inclination | 12 months
  Quantitative assessment of molars inclination between the two groups as measured by tomographic superimposition at the end of space closure.
Canine inclination | 12 months
  Quantitative assessment of canines inclination between the two groups as measured by tomographic superimposition at the end of space closure.
Incisors inclination | 12 months
  Quantitative assessment of incisors inclination between the two groups as measured by tomographic superimposition at the end of space closure.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Caetano, MSc, Principal Investigator — Rio de Janeiro State University; Flavia Artese, PhD, Study Director — Rio de Janeiro State University; Jose Augusto M Miguel, PhD, Study Chair — Rio de Janeiro State University
Locations (1):
- Faculdade de Odontologia - UERJ, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Heo W, Nahm DS, Baek SH. En masse retraction and two-step retraction of maxillary anterior teeth in adult Class I women. A comparison of anchorage loss. Angle Orthod. 2007 Nov;77(6):973-8. doi: 10.2319/111706-464.1. PMID 18004930
- [Background] Xu TM, Zhang X, Oh HS, Boyd RL, Korn EL, Baumrind S. Randomized clinical trial comparing control of maxillary anchorage with 2 retraction techniques. Am J Orthod Dentofacial Orthop. 2010 Nov;138(5):544.e1-9; discussion 544-5. doi: 10.1016/j.ajodo.2009.12.027. PMID 21055588
- [Background] Schneider PP, Gandini Junior LG, Monini ADC, Pinto ADS, Kim KB. Comparison of anterior retraction and anchorage control between en masse retraction and two-step retraction: A randomized prospective clinical trial. Angle Orthod. 2019 Mar;89(2):190-199. doi: 10.2319/051518-363.1. Epub 2018 Nov 26. PMID 30475647
- [Background] Leonardi R, Annunziata A, Licciardello V, Barbato E. Soft tissue changes following the extraction of premolars in nongrowing patients with bimaxillary protrusion. A systematic review. Angle Orthod. 2010 Jan;80(1):211-6. doi: 10.2319/010709-16.1. PMID 19852663
- [Background] Kojima Y, Fukui H. Numerical simulation of canine retraction by sliding mechanics. Am J Orthod Dentofacial Orthop. 2005 May;127(5):542-51. doi: 10.1016/j.ajodo.2004.12.007. PMID 15877034
- [Background] Bennett JC, McLaughlin RP. Controlled space closure with a preadjusted appliance system. J Clin Orthod. 1990 Apr;24(4):251-60. No abstract available. PMID 2094736
- [Background] Ribeiro GL, Jacob HB. Understanding the basis of space closure in Orthodontics for a more efficient orthodontic treatment. Dental Press J Orthod. 2016 Mar-Apr;21(2):115-25. doi: 10.1590/2177-6709.21.2.115-125.sar. PMID 27275623
- [Background] Pervin S, Rolland S, Taylor G. En masse versus two-step retraction of the anterior segment. Evid Based Dent. 2018 Dec;19(4):111-112. doi: 10.1038/sj.ebd.6401343. PMID 30573856
- [Background] Rizk MZ, Mohammed H, Ismael O, Bearn DR. Effectiveness of en masse versus two-step retraction: a systematic review and meta-analysis. Prog Orthod. 2018 Jan 5;18(1):41. doi: 10.1186/s40510-017-0196-7. PMID 29302879
- [Background] Cevidanes LH, Bailey LJ, Tucker GR Jr, Styner MA, Mol A, Phillips CL, Proffit WR, Turvey T. Superimposition of 3D cone-beam CT models of orthognathic surgery patients. Dentomaxillofac Radiol. 2005 Nov;34(6):369-75. doi: 10.1259/dmfr/17102411. PMID 16227481
- [Background] Cevidanes LH, Styner MA, Proffit WR. Image analysis and superimposition of 3-dimensional cone-beam computed tomography models. Am J Orthod Dentofacial Orthop. 2006 May;129(5):611-8. doi: 10.1016/j.ajodo.2005.12.008. PMID 16679201
- [Background] Feldmann I, Bondemark L. Orthodontic anchorage: a systematic review. Angle Orthod. 2006 May;76(3):493-501. doi: 10.1043/0003-3219(2006)076[0493:OA]2.0.CO;2. PMID 16637733
- [Background] Geron S, Shpack N, Kandos S, Davidovitch M, Vardimon AD. Anchorage loss--a multifactorial response. Angle Orthod. 2003 Dec;73(6):730-7. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 14719740
- [Background] Domingo-Clerigues M, Montiel-Company JM, Almerich-Silla JM, Garcia-Sanz V, Paredes-Gallardo V, Bellot-Arcis C. Changes in the alveolar bone thickness of maxillary incisors after orthodontic treatment involving extractions - A systematic review and meta-analysis. J Clin Exp Dent. 2019 Jan 1;11(1):e76-e84. doi: 10.4317/jced.55434. eCollection 2019 Jan. PMID 30697398
- [Background] Keim RG. Space closure and anchorage control. J Clin Orthod. 2013 Mar;47(3):153-4. No abstract available. PMID 23660788
- [Background] Keim RG. The challenge of bimaxillary protrusion. J Clin Orthod. 2017 Jun;51(6):315-316. No abstract available. PMID 29059058
- [Background] Liu Y, Olszewski R, Alexandroni ES, Enciso R, Xu T, Mah JK. The validity of in vivo tooth volume determinations from cone-beam computed tomography. Angle Orthod. 2010 Jan;80(1):160-6. doi: 10.2319/121608-639.1. PMID 19852656
- [Background] Shearn BN, Woods MG. An occlusal and cephalometric analysis of lower first and second premolar extraction effects. Am J Orthod Dentofacial Orthop. 2000 Mar;117(3):351-61. doi: 10.1016/s0889-5406(00)70240-x. PMID 10715095
- [Background] Ong HB, Woods MG. An occlusal and cephalometric analysis of maxillary first and second premolar extraction effects. Angle Orthod. 2001 Apr;71(2):90-102. doi: 10.1043/0003-3219(2001)0712.0.CO;2. PMID 11302594
- [Background] Solem RC, Marasco R, Guiterrez-Pulido L, Nielsen I, Kim SH, Nelson G. Three-dimensional soft-tissue and hard-tissue changes in the treatment of bimaxillary protrusion. Am J Orthod Dentofacial Orthop. 2013 Aug;144(2):218-28. doi: 10.1016/j.ajodo.2013.03.018. PMID 23910203
- [Background] Williams R, Hosila FJ. The effect of different extraction sites upon incisor retraction. Am J Orthod. 1976 Apr;69(4):388-410. doi: 10.1016/0002-9416(76)90208-6. PMID 1062936
- [Background] Yoshida N, Koga Y, Mimaki N, Kobayashi K. In vivo determination of the centres of resistance of maxillary anterior teeth subjected to retraction forces. Eur J Orthod. 2001 Oct;23(5):529-34. doi: 10.1093/ejo/23.5.529. PMID 11668872